CLINICAL TRIAL: NCT03007771
Title: A Feasibility Study of Magnetic Resonance-guided High-Intensity Focused Ultrasound (MR-HIFU) Used for Mild Hyperthermia in Human Subjects
Brief Title: Magnetic Resonance-guided High-Intensity Focused Ultrasound (MR-HIFU) Used for Mild Hyperthermia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Decision was made to not go forward with the study
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 201612155
Record Dates: First submitted 2016-12-29; First posted 2017-01-02 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Healthy Participants; Pelvic Neoplasms; Soft-tissue Sarcoma; Bladder Cancer; Cervical Cancer; Rectal Cancer
MeSH Terms: conditions — Pelvic Neoplasms; Sarcoma; Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- MR-HIFU (Experimental): * Philips 1.5T MRI scanner equipped with a Sonalleve V2 HIFU system will be used
  * Will be scanned in the MRI in 1 or more positions to the extremities and/or pelvis while aligned to the HIFU system. The HIFU device will then be used to apply sub-clinical levels (≤ 41°C) of heat to one or more small volumes. Regions will be heated to the desired temperature for variable short durations of time not exceeding 30 minutes.
  * After the session is complete, the patient will be removed from the MR-HIFU system and, following a 15-30-minute period of monitoring for any adverse events, allowed to leave.
  * Before the scan, after the scan and 5-10 days following the scan, participants will be asked to rate any pain, discomfort, in the area to be heated, as well as any anxiety or claustrophobia on a scale of 1-10 with 1 being minimal/none and 10 being extreme. The skin area to be treated will also be reviewed for any redness/discoloration.
  Interventions: Device: Magnetic Resonance-guided High-Intensity Focused Ultrasound

INTERVENTIONS:
Device: Magnetic Resonance-guided High-Intensity Focused Ultrasound — -Heating will not be performed in two areas of the body near each other (for example, not heating in two different places of the same thigh) to minimize the risk of overheating any one part of the subject's body. Heating a second target site is not mandatory, even if time allows, and the participant may refuse.
  Other Names: MR-HIFU

SUMMARY:
This study will help to elucidate the treatment sites in the extremities and pelvis for which MR-guided HIFU heating is feasible, which has the potential to be beneficial for patients with conditions at those sites (soft tissue sarcoma, cervical cancer, etc.). The investigators anticipate that successful completion of this study will lead to clinical trials in those feasible sites of interest to determine the safety and efficacy of administering therapeutic levels of heat for hyperthermia or other applications.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Willing and able to provide informed consent
* Patients only: must have a tumor in extremity muscle tissue or in the pelvis.

Exclusion Criteria:

* Contraindications for MRI (e.g., unsafe MRI implanted devices, shrapnel, history of metal fragments in eyes, neurostimulators, excessive size and weight, claustrophobia)
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-30 (Estimated); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the MR-HIFU device as measured by whether an area can be heated to the designated temperature and held at that temperature for an appropriate time frame | 1 day (2 hour timeframe)
  -Temperature in the participant will be monitored using MR thermometry with the MR scanner
Feasibility of the MR-HIFU device as measured by whether an area can be heated while simultaneously maintaining patient comfort | Up to 10 days
  * Patient comfort will be measured by the Comfort Score. Before the scan, participants will be asked to rate any pain, discomfort, in the area to be heated, as well as any anxiety or claustrophobia on a scale of 1-10 with 1 being minimal/none and 10 being extreme. The skin area to be treated will also be reviewed for any redness/discoloration. After the scan, the same questions will be asked again of the subject.
  * Participants will be contacted by phone 5-10 days following participation in the study. Participants will be asked to describe any negative effects in the area heated since participation in the study, including pain, discomfort, and/or cosmetic changes (such as skin redness). Participants will be asked to score pain/discomfort on a scale of 1-10, with 1 being minimal/none and 10 being extreme.
Feasibility of the MR-HIFU device as measured by whether coupling can be maintained with the body area in the same position while having contact with the transducer for an appropriate time frame. | 1 day (2 hour timeframe)
  -Patients' skin will be cooled using the MR-HIFU system's direct skin cooling device to minimize over heating of the skin, unless one or more gel pads are required to achieve proper coupling to the HIFU system. In order to ensure good contact with the surface of the HIFU interface, participants may be shaved or have other hair-removal products applied to limited regions of their body.

SECONDARY OUTCOMES:
Behavior of hyperthermia delivery as measured by the build-up of time until the different treatment cells can reach a desired uniform temperature | 1 day (2 hour time frame)
  --Temperature in the participant will be monitored using MR thermometry with the MR scanner
Behavior of hyperthermia delivery as measured by if the heating cell behavior is the same in healthy and tumor tissues | 1 day (2 hour time frame)
  --Temperature in the participant will be monitored using MR thermometry with the MR scanner
Behavior of hyperthermia delivery as measured by post-treatment heat diffusion behavior to anticipate any issues when heat is given at a clinically relevant level | Up to 10 days
  -Participants will be contacted by phone 5-10 days following participation in the study. Participants will be asked to describe any negative effects in the area heated since participation in the study, including pain, discomfort, and/or cosmetic changes (such as skin redness).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Altman, Ph.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu